CLINICAL TRIAL: NCT06188494
Title: A Multicenter, Observational, Secondary Data Collection, Retrospective, National Study to Assess the Prevalence of HER2-low Breast Cancer Among Patients Previously Diagnosed With Unresectable and/or Metastatic HER2-Negative Breast Cancer in Egypt - UNFOLD
Brief Title: UNFOLD Study Egypt
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D133FR00199
Record Dates: First submitted 2023-11-13; First posted 2024-01-03 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Breast cancer is a major public health concern worldwide. In Egypt, it was the most diagnosed cancer among females in 2020 with an incidence rate of 32.4%. Its age-standardized incidence and mortality rates were 48.7 and 20.4 per 100,000 population, respectively. The status quo of HER2 testing in Egypt is that all breast cancer cases are tested for HER2 protein expression on the surface of tumor cells by immunohistochemistry (IHC), and only those with score 2 (equivocal) and selected cases of score 3 are subjected for further analysis using in-situ hybridization technique (ISH) to detect HER2 gene amplification in tumor nuclei.

DETAILED DESCRIPTION:
Besides its role in the prognostic assessment of breast cancer, accurate determination of HER2 status is critical for appropriate selection of eligible patients for targeted therapy. In 2018, the American Society of Clinical Oncology (ASCO) and the College of American Pathologists (CAP) had a revised guideline for HER2 testing in breast cancer. Breast cancers were traditionally classified as HER2-pos and HER2-neg. HER2-positive BCs are those with either IHC3+ -characterized as complete, intense circumferential membrane staining in >10% of cells-, or equivocal IHC (i.e., IHC2+) -characterized as weak to moderate/complete membrane staining in >10% of cells- and ISH+. While HER2-negative BCs were considered those with one of the following results: IHC0 (No staining or incomplete, faint/barely perceptible staining in ≤10% of cells), IHC1+ (No staining or incomplete, faint/barely perceptible staining in >10% of cells), or IHC2+ and ISH-. Recently, the HER2 categorization of BC has been differentiated into 3 subgroups: those with no detectable IHC staining (referred to herein as HER2 null), those with detectable HER2 staining in less than 10% of tumor cells (referred to herein as IHC>0<1+), and those with IHC1+ or IHC2+/ISH- results (collectively referred to herein as HER2-low). Little is known about the prevalence and clinical implications of HER2-neg BC subgroups that express low levels of HER2; these cancers have traditionally not been considered as separate subgroups and consequently there has been a lack of HER2-directed treatment options for these patients.

Treatment options for mBC depend on several factors including, but not limited to, the patient's overall health and the levels of hormone receptor (HR) and HER2 in the tumor. Current SoC that is based on HER2 expression only considers BCs as being either HER2-pos or HER2-neg. For HER2-pos cancers, therapies that target HER2 combined with chemotherapy or other anti-HER2 agents can significantly improve survival. Although there are no therapies specifically for patients with HER2-low BC, preliminary evidence has demonstrated antitumor activity of T-DXd, an anti-HER2 agent, in HER2-low BCs. Hence, applying the most recent cut-off values when testing for HER2 expression is critical for maximizing treatment benefit for the highest number of patients (HER2-low & HER2-pos).

This national, multicenter, non-interventional, secondary data collection, retrospective study aims to describe the prevalence of HER2-low BC in Egypt by accurate categorization of HER2 status in HER2 reports of patients previously determined as HER2-neg and analyzing the SoC and clinical outcomes of HER2-low patients from medical chart abstraction.

ELIGIBILITY:
Inclusion Criteria:

1. Men or women ≥ 18 years of age,
2. Must have a histological, cytological, or radiological confirmed diagnosis of unresectable or/and mBC between 01 January 2017 and 31 December 2020, with at least 2 years of follow-up data unless patient's death is confirmed,
3. Diagnosed as HER2-neg (HER2 IHC 0, 1+, 2+/ISH-), regardless of hormone status,
4. Must have a report in her file with HER2 scoring with IHC/ISH or both,
5. Progressed on any systemic anti-cancer therapy (eg, ET, chemotherapy, CDK4/6i, targeted therapies other than anti-HER2, or immunotherapy) in the metastatic setting.
6. Due to the retrospective nature of the study a waiver grant of the consent will be requested from the IRB/IEC for the study participants, if waiver not granted Patient or next of kin/legal representative (for deceased patients at study entry) willing and able to provide written informed consent according to the local regulations.

Exclusion Criteria:

* Records of patients who meet any of the following criteria will be excluded:

  1. History of other malignancies than mBC,
  2. Historical HER2 status of IHC 2+/ISH+ or 3+, or HER2 amplified.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with confirmed diagnosis of HER2-negative, unresectable and/or mBC (regardless of HR status) between 01 January 2017 and 31 December 2020 who progressed on any systematic anticancer therapy (eg, ET, chemotherapy, CDK4/6i, targeted therapies other than anti-HER2, or immunotherapy). Patients' clinical outcomes will be followed up for 2 years after the date of their diagnosis.
Sampling Method: Non-Probability Sample
Enrollment: 405 (Actual)
Dates: Start 2024-05-13 (Actual); Primary Completion 2024-09-16 (Actual); Study Completion 2024-09-16 (Actual)

PRIMARY OUTCOMES:
HER2-low prevalence | 3 Years
  HER2-low prevalence based on reviewing historical HER2 reports of HER2-neg mBC patients.

SECONDARY OUTCOMES:
HER2-low Breast Cancer Patient Baseline characteristics | 3 Years
  Baseline characteristics for patients identified as having HER2-low BC.
HER2 IHC Null Breast Cancer Patient Baseline Characteristics | 3 Years
  Baseline characteristics for patients identified as having HER2 IHC Null BC.
The overall prevalence of HER2-low among unresectable and/or mBC patients | 3 Years
  The overall prevalence of HER2-low among unresectable and/or mBC patients identified as HER2-neg, regardless of assays used, will also be summarized descriptively for HR-pos and HR-neg population, respectively.
Treatment patterns | 3 Years
  Types of therapies for patients will be summarized descriptively for HR-pos and HR-neg population, respectively.
HER2-low Breast Cancer Clinical presentation for patients | 3 Years
  clinical presentation for patients identified as having HER2-low BC.
HER2 IHC Null Breast Cancer clinical presentation for patients | 3 Years
  clinical presentation for patients identified as having HER2 IHC Null BC.
HER2-low Breast Cancer Patients Clinical outcomes | 3 Years
  Clinical outcomes for patients identified as having HER2-low BC.
HER2 IHC Null Breast Cancer Patients Clinical outcome | 3 Years
  Clinical outcomes for patients identified as having HER2 IHC Null BC.
Treatment Patterns | 3 Years
  Duration on treatment therapies for patients will be summarized descriptively for HR-pos and HR-neg population, respectively.

CONTACTS AND LOCATIONS:
Locations (7):
- Egypt (7):
  - Research Site, Alexandria
  - Research Site, Asyut
  - Research Site, Cairo
  - Research Site, Gharbia
  - Research Site, Giza
  - Research Site, Luxor
  - Research Site, Sohag

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: CSR Synopsis redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D133FR00199&attachmentIdentifier=167280a9-7f3b-42db-9574-95e13537c662&fileName=CSR_Synopsis_redacted.pdf&versionIdentifier=